CLINICAL TRIAL: NCT03895021
Title: "Stepping On" to Pisando Fuerte: Adapting an Evidence-Based Falls Prevention Program for Latino Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United Community Center (Other); Centro Hispano (Unknown); North/Eastside Senior Coalition (Unknown); Latino Health Council (Unknown); Greater Wisconsin Agency on Aging Resources (Unknown); Community-Academic Aging Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-1311
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Falls Prevention
Keywords: falls prevention; Latino; Hispanic; Stepping On

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This multifaceted, adapted program focuses preventing falls through balance and strength exercises, teachings from guest experts (e.g., PT, Pharmacist, vision) and at-home safety education. Participants attended weekly 2-hour group sessions (8 -12 persons) over the course of 8 weeks delivered in Spanish by trained Hispanic/Latino personnel in two communities in Wisconsin.
  Interventions: Behavioral: Pisando Fuerte

INTERVENTIONS:
Behavioral: Pisando Fuerte — "Pisando Fuerte", a linguistically and culturally appropriate version for Spanish speakers of an evidence-based fall prevention program ("Stepping On" [SO]).

SUMMARY:
There are no evidence-based fall prevention programs for Hispanic/Latinos even though their age-adjusted death rate from unintentional falls is climbing in the US. "Pisando Fuerte", a linguistically and culturally appropriate version of an evidence-based fall prevention program for Spanish speakers ("Stepping On" [SO]) is evaluated. "Pisando Fuerte" consists of 2-hour group sessions over the course of 8 weeks delivered in Spanish by trained Hispanic/Latino personnel in two communities in Wisconsin. Implementation and intervention fidelity were evaluated by an independent assessor on three sessions using a-priori criteria based on key elements of SO. Uptake, proximal and distal outcomes were assessed through interviews 6 months after the program.

DETAILED DESCRIPTION:
Stepping On is an evidence-based falls prevention program for community-dwelling persons 65+. It uses principles of self-efficacy in 2-hour sessions held once a week for 7 weeks + one home visit to review principles learned in class and one booster class after 3 months.

The program, developed and researched in Australia, was found to reduce falls by 30%. It was brought to the U.S. in 2006 by the Kenosha County Aging Division in collaboration with Dr. Jane Mahoney, U.W. Madison and other Wisconsin partners using foundation and state funding. Funding from the CDC provided the opportunity to adapt the program for widespread dissemination in the United States. In addition preliminary work was done on translating and culturally adapting Stepping On for the Latino community. The adapted program, known as Pisando, was offered as a pilot class at the United Community Center in Milwaukee in 2012. Further revisions were made to the program based on the experience at the pilot classes and advice from the advisory board, but questions remained about some key areas of workshop format.

ELIGIBILITY:
Inclusion Criteria:

- Have fallen in the past year

Exclusion Criteria:

* Living arrangement does not include a kitchen of their own (i.e., independent living)
* Unable to walk without help from another person, ambulate independently
* Reliant on a walker to get around inside of home

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Falls per person | 6 months
  To help test effectiveness; direct empirical evidence. Results will be reported as an average number.
Falls Behavioral Scale (FaB) | 6 months
  To help test implementation; direct empirical evidence. Shortened Fall Behavioral Scale (FaB) scale, a 24-item validated tool that assesses the presence of protective behaviors for falls in older adults using a scale between 0 (not at all) and 4 (very much). High scores indicate the safest behaviors and low scores indicate risky behaviors. Total averaged scores range from 1-4.
Fidelity of Enactment | 1 week and 6 months
  To help test implementation; proxy empirical evidence. This is an assessment of fidelity of participants' whom engaged in intermediary falls prevention behaviors after Pisando Fuerte ended (two time-points: at 1-week post-intervention and 6 months post-intervention), expressed as a percentage. Falls prevention behavior measures include: exercise adherence, elimination of at-home falls hazards, and adjustments to walking form and standing posture.
Fidelity of delivery | 6 months
  To help test implementation; direct empirical evidence. This is an assessment of fidelity of trained Pisando Fuerte leaders' delivery of the program's key elements (as determined in the original Stepping On program), expressed as a percentage for each component/element. Elements measured for fidelity of delivery include: Adult Learning, Program Aspects, Exercise Element, Upgrading Exercise, Background & Training of Group Leader, Group Leader's Role, Elements of Peer Co-leader Role, and Cultural Adaption (specific to Pisando Fuerte, not included in Stepping On). The benchmark to be considered sufficient fidelity of delivery is 80%.
Reach | 6 months
  Number of individuals screened, enrolled, completed program; direct empirical evidence
Timed Up and Go (TUG) | Up to 8 weeks
  Assess mobility, balance, walking ability and fall risk in older adults. Assessors used the following instruction: "Levantese de la silla, camine 10 pies a un paso cómodo, gire, y regrese a la silla a sentarse otra vez", which translates to: "Stand up from the chair, walk 10 feet using a comfortable pace, turn around, and walk back and sit down." An older adult who takes 12+ seconds to complete is considered at risk for falling.

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Mahoney, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - North/Eastside Senior Coalition (NewBridge Madison), Madison, Wisconsin
  - Centro Hispano, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aarons GA, Sklar M, Mustanski B, Benbow N, Brown CH. "Scaling-out" evidence-based interventions to new populations or new health care delivery systems. Implement Sci. 2017 Sep 6;12(1):111. doi: 10.1186/s13012-017-0640-6. PMID 28877746
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Ford JH 2nd, Abramson B, Wise M, Dattalo M, Mahoney JE. Bringing Healthy Aging to Scale: A Randomized Trial of a Quality Improvement Intervention to Increase Adoption of Evidence-Based Health Promotion Programs by Community Partners. J Public Health Manag Pract. 2017 Sep/Oct;23(5):e17-e24. doi: 10.1097/PHH.0000000000000503. PMID 27997482
- [Background] Mahoney JE, Clemson L, Schlotthauer A, Mack KA, Shea T, Gobel V, Cech S. Modified Delphi Consensus to Suggest Key Elements of Stepping On Falls Prevention Program. Front Public Health. 2017 Feb 20;5:21. doi: 10.3389/fpubh.2017.00021. eCollection 2017. PMID 28265557
- [Derived] Mora Pinzon M, Myers S, Jacobs EA, Ohly S, Bonet-Vazquez M, Villa M, Castro A, Mahoney J. "Pisando Fuerte": an evidence-based falls prevention program for Hispanic/Latinos older adults: results of an implementation trial. BMC Geriatr. 2019 Sep 18;19(1):258. doi: 10.1186/s12877-019-1273-1. PMID 31533636